CLINICAL TRIAL: NCT06373523
Title: MASLD in Primary Hypothyroidism and Efficacy of Dapaglifozin
Acronym: SHIELD
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Ashu Rastogi, Associate Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHIELD
Record Dates: First submitted 2023-12-17; First posted 2024-04-18 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Hepatic Steato-Fibrosis; Non-Alcoholic Fatty Liver Disease
Keywords: Dapaglifozin; MRI-PDFF; Primary hypothyroidism
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Hypothyroidism | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: Eligible subjects will be randomly allocated to either the Dapagliflozin group or placebo group (i.e. control group)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The placebo pills will be manufactured in identical appearance to the study drug (Dapagliflozin)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dapagliflozin Plus levothyroxine Group (Experimental): Dapagliflozin 10mg daily will be given to the treatment arm in addition to Levothyroxine replacement therapy. Eligible subjects will be followed up until week 28, and will undergo clinical, anthropometric and laboratory assessments (including liver function test and lipid profile) at baseline, week 14 and week 28. They will undergo LSM and CAP By Transient Elastography at baseline, week 14 and week 28, and MRI-PDFF at baseline and week 28. The primary outcome will be a difference in change of liver fat content (measured by MRI-PDFF) at week 28 from baseline between the two groups. The secondary outcomes will be proportion of participants achieving remission of steatosis (MRIPDFF <5%) at week 28, reduction of liver fibrosis (LSM) and decrease in hepatic steatosis by 1 stage at week 14 and 28 and other secondary outcomes as mentioned above.
  Interventions: Drug: Dapagliflozin 10mg Tab; Drug: Levothyroxine Replacement daily
- Levothyroxine daily and Placebo pill identical to Dapaglifozin for 28 weeks (Placebo Comparator): The placebo pill will be manufactured to identical in appearance to the Dapaglifozin will be given to the Placebo arm in addition to Levothyroxine replacement therapy. Eligible subjects will be followed up until week 28, and will undergo clinical, anthropometric and laboratory assessments (including liver function test and lipid profile) at baseline, week 14 and week 28. They will undergo LSM and CAP By Transient Elastography at baseline, week 14 and week 28, and MRI-PDFF at baseline and week 28. The primary outcome will be a difference in change of liver fat content (measured by MRI-PDFF) at week 28 from baseline between the two groups. The secondary outcomes will be proportion of participants achieving remission of steatosis (MRI PDFF <5%) at week 28, reduction of liver fibrosis (LSM) and decrease in hepatic steatosis by 1 stage at week 14 and 28 and other secondary outcomes as mentioned above.
  Interventions: Drug: Placebo; Drug: Levothyroxine Replacement daily

INTERVENTIONS:
Drug: Dapagliflozin 10mg Tab — Dapagliflozin 10mg daily will be given to the treatment arm.Eligible subjects will be followed up until week 28, and will undergo clinical, anthropometric and laboratory assessments (including liver function test and lipid profile) at baseline, week 14 and week 28. They will undergo LSM and CAP By Transient Elastography at baseline, week 14 and week 28, and MRI-PDFF at baseline and week 28. The primary outcome will be a difference in change of liver fat content (measured by MRI-PDFF) at week 28 from baseline between the two groups.
  Other Names: Dartdapa
  Arms: Dapagliflozin Plus levothyroxine Group
Drug: Placebo — The placebo pills will be manufactured to be identical in appearance to the study drug(Dapaglifozin 10 mg tablet).
  Other Names: Placib
  Arms: Levothyroxine daily and Placebo pill identical to Dapaglifozin for 28 weeks
Drug: Levothyroxine Replacement daily — Levothyroxine Replacement daily for 28 weeka
  Other Names: LT4

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) is a global epidemic with a prevalence of 25-40%.Primary Hypothyroidism is one of Endocrinopathies who are at risk of developing NAFLD/NASH and estimated prevalence of Primary Hypothyroidism in NAFLD patients is 10-15 %.Though First line Management is Dietary changes and lifestyle modifications(LSM),unfortunately Adherence to Lifestyle has been poor,rise of Lean NAFLD is on rise, faster progression of NAFLD,evolving risk factors for NAFLD like endocrinopathies,these push need for Pharmacotherapy.Currently therapies for NAFLD patients without diabetes mellitus (DM) are limited, and are associated with various adverse side effects. Sodium-glucose cotransporter type-2 (SGLT2) inhibitors can reduce hepatic fat content in patients with DM which is independent of glycemic control. However, the role of SGLT2 inhibitors in NAFLD patients without DM has not been investigated.Magnetic resonance imaging-derived proton density fat fraction (MRI-PDFF) is an emerging non-invasive imaging technique, and is more sensitive than liver biopsy/histology in quantifying liver fat change. Liver stiffness measurement (LSM) by Transient Elastography is a non-invasive method to diagnose fibrosis/cirrhosis with high accuracy.The novelty of utilizing the concept of "drug repositioning" by changing the role of SGLT2 inhibitors in treating DM to treating NAFLD in patients without DM deserves exploration.The investigators propose a double-blind, randomized, placebo-controlled trial to compare the effects of Dapagliflozin (a type of SLGT2 inhibitors) versus placebo (in a 1:1 ratio) in reducing hepatic fat content as measured by MRI-PDFF in NAFLD patients with Primary Hypothyroidism.The study results will determine whether SGLT2 inhibitors can reduce hepatic steatosis/hepatic fibrosis in NAFLD patients with Primary Hypothyroidism.

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) is a global epidemic with a prevalence of 25-40%.Cirrhosis can occur without intervening NASH .Time line of progression is variable - modified by risk factors.Over all average progression from one disease Stage to another can take up 7 years for NASH while 14 years for NAFLD.In general ,10-30% of patient NAFLD progress to NASH ; Of which 15-25 % progress to advanced fibrosis.Amongst advanced fibrosis,20 % Progress to Cirrhosis over 2 years and 20 % of cirrhotics will have decompensation over 2 years.Overall in NAFLD MCC of mortality - CVD>Extrahepatic cancer > Liver specific mortality ( HCC and Hepatic decompensation).Primary Hypothyroidism is one of Endocrinopathies who are at risk of developing NAFLD/NASH and estimated prevalence of Primary Hypothyroidism in NAFLD patients is 10-15 %.

Though First line Management is Dietary changes and lifestyle modifications(LSM),unfortunately Adherence to Lifestyle has been poor,rise of Lean NAFLD is on rise, faster progression of NAFLD,evolving risk factors for NAFLD like endocrinopathies,these push need for Pharmacotherapy.Currently therapies for NAFLD patients without diabetes mellitus (DM) are limited, and are associated with various adverse side effects. Sodium-glucose cotransporter type-2 (SGLT2) inhibitors can reduce hepatic fat content in patients with DM which is independent of glycemic control. However, the role of SGLT2 inhibitors in NAFLD patients without DM has not been investigated.

Magnetic resonance imaging-derived proton density fat fraction (MRI-PDFF) is an emerging non-invasive imaging technique, and is more sensitive than liver biopsy/histology in quantifying liver fat change.The Dixon proton density fat fraction sequence is frequently used to determine the liver's fat composition.To estimate PDFF across the entire liver, 9 regions of interest (ROIs) of 200 mm2 to 300 mm2 in the area will be placed in the nine liver segments on the PDFF parametric maps.This fat percentage called PDFF is calculated by the following formula; PDFF

= F / (F +W) x 100% The radiological findings will be examined by the radiology investigator who will be blinded to prior liver fat fraction maps.

Liver stiffness measurement (LSM) by Transient Elastography is a non-invasive method to diagnose fibrosis/cirrhosis with high accuracy.

The novelty of utilizing the concept of "drug repositioning" by changing the role of SGLT2 inhibitors in treating DM to treating NAFLD in patients without DM deserves exploration.

The investigators propose a double-blind, randomized, placebo-controlled trial to compare the effects of Dapagliflozin (a type of SLGT2 inhibitors) versus placebo (in a 1:1 ratio) in reducing hepatic fat content as measured by MRI-PDFF in NAFLD patients with Primary Hypothyroidism.

A total of 60 adult patients will be randomly sampled from the Endocrinology/liver/Internal Medicine clinics from our institute. Dapagliflozin 10mg daily will be given to the treatment arm. The placebo pill will be manufactured to be identical in appearance to the study drug. Eligible subjects will be followed up until week 28, and will undergo clinical, anthropometric and laboratory assessments (including Liver function test and Lipid profile) at baseline, week 4, 12 and 28 weeks. They will undergo LSM/CAP at baseline, week 14 and 28, and MRI-PDFF at baseline and week 28. The primary outcome will be a difference in change of liver fat content (measured by MRI-PDFF) at week 28 from baseline between the two groups. The secondary outcomes will be proportion of participants achieving remission of steatosis (MRI-PDFF <5%) at week 28, reduction of liver fibrosis (LSM) and decrease in steatosis by 1 stage at week 14 and 28, improvement of laboratory results (including liver transaminases and ductal enzymes, fasting glucose, HbA1c, lipid profile), improvement of anthropometric measurements, and cardiovascular events.

The study results will determine whether SGLT2 inhibitors can reduce hepatic steatosis and regress fibrosis in NAFLD patients with Primary Hypothyroidism.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years
2. Patients with Primary Overt hypothyroidism (Low FT3/Low FT4 and TSH>ULN)

Exclusion Criteria:

1. Patients with Diabetes Mellitus(T1DM AND T2DM)
2. Patient with Secondary Hypothyroidism
3. Patients with other Endocrinopathies who are at risk of MASLD (T1DM and T2DM, Growth Hormone Insufficiency,Cushing Syndrome)
4. Patients with concomitant other etiologies for hepatic steatosis or elevated transaminases (chronic viral hepatitis infection, autoimmune hepatitis, Wilson's disease, hemochromatosis, congestive hepatopathy, primary biliary cholangitis, primary sclerosing cholangitis, biliary tract obstruction)
5. Patient with Drug Induced Liver Injury(DILI)
6. Patients with Decompensated Cirrhosis or Portal hypertensionPatients with Cirrhosis or Portal hypertension
7. Patients with HCC or any other malignancy
8. Drugs like OCPS
9. Patients <18 years of age
10. Patients already on Vitamin E or pioglitazone
11. Pregnancy/Lactation
12. Patients who are too sick to carry out the protocol
13. Those who do not consent to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Change in liver fat content | 28 weeks
  Difference in the change in liver fat content between the two groups at week 28 from the baseline as measured by MRI-PDFF

SECONDARY OUTCOMES:
Proportion of participants achieving 1 Stage decrease in steatosis at 6 months asassessed by Transient Elastography | 28 weeks
  Proportion of participants achieving 1 Stage decrease in steatosis at 6 months as assessed by Transient Elastography
Changes in Improvement in hepatic fibrosis measured by non invasive parameters like Fib4 score at 3 and 6 months | 28 weeks
  Changes in Improvement in hepatic fibrosis measured by non invasive parameters like Fib4 score at 3 and 6 months
Changes in Lipid Profile at 3 and 6 months | 28 weeks
  Changes in Lipid Profile at 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ashu Rastogi, MD,DM, Principal Investigator — PGIMER, Chandigarh
Locations (1):
- PGIMER, Chandigarh, Punjab, India

IPD SHARING:
Plan to Share IPD: No